CLINICAL TRIAL: NCT04667234
Title: A Multicenter, Open-label, Single-arm, Expanded Access Protocol of Sotorasib for the Treatment of Subjects With Previously Treated Locally Advanced Unresectable/Metastatic NSCLC With KRAS p.G12C Mutation
Brief Title: Expanded Access of Sotorasib
Status: No longer available | Type: Expanded Access
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20190436
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Non Small-cell Lung Cancer; Locally Advanced Unresectable NSCLC; Locally Advanced Metastatic NSCLC
Keywords: NSCLC; KRAS p.G12C Mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sotorasib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: AMG 510 — Administered as an oral tablet.
  Other Names: Sotorasib; Lumakras (US); Lumykras (UK)

SUMMARY:
The primary objective of this study is to provide expanded access to and characterize the safety profile of Sotorasib in participants with previously treated locally advanced/unresectable/metastatic non small-cell lung cancer (NSCLC) with KRAS p.G12C mutation in a real-world setting.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years
* Ineligibility for participation in any Amgen-sponsored ongoing clinical study of the investigational product
* Pathologically documented, locally-advanced and unresectable or metastatic Non Small-Cell Lung Cancer (NSCLC) with KRAS p.G12C mutation confirmed through molecular testing
* Exhausted other standard of care options for locally advanced and unresectable or metastatic NSCLC disease including platinum-based combination chemotherapy and programmed cell death protein 1/programmed death-ligand 1 (PD 1/PD-L1) immunotherapy (unless medically contraindicated)
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2

Exclusion Criteria

* Mixed small-cell lung cancer or mixed NSCLC histology
* Active brain metastases
* Active hepatitis B or hepatitis C virus
* Current active malignancy other than NSCLC
* Currently or previously enrolled in a prior sotorasib study unless radiographic disease progression confirmed, able to remain on long term follow up of their original protocol and receives medical monitor approval
* Female participants planning to become pregnant while on study through 7 days after the last dose of sotorasib

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (55):
- United States (30):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Ironwood Cancer and Research Center, Chandler, Arizona
  - Arizona Oncology Associates Professional Corporation, Tucson, Arizona
  - San Luis Valley Health Regional Medical Center, Alamosa, Colorado
  - Kaiser Permanente, Lone Tree, Colorado
  - Sacred Heart Medical Oncology Group, Pensacola, Florida
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - McFarland Clinic PC, Ames, Iowa
  - Des Moines Oncology Research Association, Des Moines, Iowa
  - Saint Joseph East, Lexington, Kentucky
  - Louisiana Hematology Oncology Associates, Baton Rouge, Louisiana
  - Northern Light Cancer Center, Brewer, Maine
  - University of Pittsburgh Medical Center Western Maryland, Cumberland, Maryland
  - Maryland Oncology Hematology, PA, Rockville, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mid Michigan Medical Center, Midland, Michigan
  - Saint Lukes Cancer Institute, Kansas City, Missouri
  - Oncology Hematology Associates, Springfield, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - Wake Forest Baptist Comprehensive Cancer Research Center, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Institute, Cleveland, Ohio
  - LeHigh Valley Hospital, Allentown, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Erlanger East Hospital, Chattanooga, Tennessee
  - Baptist Cancer Center, Memphis, Tennessee
  - Saint Marys Medical Center, Huntington, West Virginia
- Argentina (4):
  - Instituto Médico Especializado Alexander Fleming, Capital Federal, Buenos Aires
  - Hospital Aleman, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Cemic, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Clínica Universitaria Privada Reina Fabiola, Córdoba
- Brazil (7):
  - Hospital Sirio Libanes, Brasília, Federal District
  - Personal Oncologia de Precisao e Personalizada, Belo Horizonte, Minas Gerais
  - Instituto de Oncologia do Parana, Curitiba, Paraná
  - Liga Norte-Riograndense Contra O Cancer, Natal, Rio Grande do Norte
  - YNOVA Pesquisa Clinica, Florianópolis, Santa Catarina
  - Fundacao Pio 12 Hospital de Cancer de Barretos, Barretos, São Paulo
  - Oncoclinicas Rio de Janeiro S A, Rio de Janeiro/RJ
- Israel (3):
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Shaare Zedek Medical Center, Petah Tikva
- Saudi Arabia (4):
  - King Fahad Specialist Hospital, Dammam
  - King Abdulaziz Medical City - National Guard Hospital, Riyadh
  - King Saud University Medical City-King Khalid University Hospital, Riyadh
  - King Faisal Specialist Hospital, Riyadh
- Taiwan (7):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Veterans General Hospital - Taichung, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com